CLINICAL TRIAL: NCT06329518
Title: Pharmacokinetics and Ex Vivo Sequestration of Rezafungin in Critically Ill Patients Receiving Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Rezafungin Pharmacokinetics in Patients on ECMO
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI departure
Sponsor: Hartford Hospital (Other)
Collaborators: Melinta Therapeutics, LLC (Industry)
Responsible Party: Principal Investigator, Joseph L. Kuti, PharmD, Director, Center for Anti-Infective Research and Development, Hartford Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HHC-2024-0064
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Sepsis
Keywords: pharmacokinetics; echinocandins
MeSH Terms: conditions — Sepsis | interventions — Rezafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rezafungin (Experimental): Participants will receive one dose of rezafungin as per current prescribing information.
  Interventions: Drug: Rezafungin

INTERVENTIONS:
Drug: Rezafungin — After receipt of Rezafungin, blood samples will be collected at various time points to determine the pharmacokinetics of Rezafungin.
  Other Names: rezafungin acetate

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a form of cardiopulmonary life-support for critically ill patients where blood is extracted from the vascular system and circulated by a mechanical pump while it is oxygenated and reinfused into the patient's circulation. It is well known that critically ill patients may experience alterations in antibiotic pharmacokinetics, and as a result, dosing modifications are generally required. There is a need to understand how ECMO circuits affect the pharmacokinetics and disposition of drugs. This study is designed to assess the pharmacokinetics of the new broad-spectrum echinocandin, Rezafungin, in critically ill patients receiving ECMO

DETAILED DESCRIPTION:
This is a prospective, open-label, Phase 1b, pharmacokinetic study of Rezafungin in 8 critically ill patients receiving ECMO support at Hartford Hospital. Informed consent will be collected from all study participants, legal authorized representative, or their next of kin in order to participate. This is not a treatment study; all participants will receive other antibiotics as necessary to treat any current infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receiving venovenous or venoarterial ECMO support.

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* History of any moderate or severe hypersensitivity or allergic reaction to any echinocandin antifungal
* Receiving rezafungin to treat documented or suspected infection within 14 days of screening, or expected to receive rezafungin during the study intervention phase
* Receiving or likely to require intermittent hemodialysis
* A hemoglobin less than 7.2 gm/dl at baseline
* Acute liver injury, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal, or AST or ALT > 3 times the upper limit of normal with an associated total bilirubin > 2 times upper limit of normal
* Patients expected to have ECMO discontinued within the next 24 hours
* Any rapidly progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)
* Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Rezafungin Clearance | 168 hours
  The Clearance in liters/hour of Rezafungin from the plasma of critically ill patients receiving ECMO

SECONDARY OUTCOMES:
Rezafungin Area Under the Curve (AUC) | 168 hours
  The AUC in milligram*hour/liter of Rezafungin calculated from concentrations collected between zero and 168 hours at steady-state.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L. Kuti, PharmD, Principal Investigator — Hartford Hospital